CLINICAL TRIAL: NCT06966531
Title: Prevalence of Myocarditis in Patients Suspected Myocardial Infarction With Non-Obstructive Coronary Arteries
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Thabit Mohamed, Resident , department of Cardiology،Principal Investigator, Assiut University
Other Study IDs: Myocarditis in MINOCA
Record Dates: First submitted 2025-05-04; First posted 2025-05-12 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Prevalence of Myocarditis in MINOCA Patients
Keywords: Myocarditis; MINOCA; Normal coronary angiography
MeSH Terms: conditions — Myocarditis; MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MINOCA: Acute Myocardial infarction patient with non obstructive coronary arteries
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography — distinguish between true MI with significant lesion and MINOCA with insignificant lesions (less than 50%)

SUMMARY:
This study aims to determine the prevalence of myocarditis among patients suspected of having myocardial infarction with non-obstructive coronary arteries (MINOCA) and to analyze its clinical characteristics, diagnostic markers .

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) remains the leading causes of high morbidity and mortality worldwide, Recently, a distinct population with myocardial infarction with nonobstructive coronary arteries (MINOCA) has been increasingly recognized because of the widespread use of coronary angiography. MINOCA occurs in 5%-10% of all AMI and they are younger and more often women compared to patients with AMI and obstructive coronary artery disease (CAD) , The underlying causes of MINOCA are manifold and may include plaque rupture or erosion, thromboembolism, coronary spasm, spontaneous dissection, microvascular dysfunction and supply/demand mismatch. Some non-ischemic diseases such as myocarditis may also mimic the presentation of MINOCA .Of note, several studies have found that the prognosis of MINOCA is not trivial and patients are still at considerable risks for long-term adverse cardiovascular (CV) events despite the optimal secondary prevention treatments [[6], [7], [8], [9], [10]]. Thus, it is of necessity and profound implications to find potential residual risk factors and improve prognosis in MINOCA population.

Myocarditis is commonly caused by viral infections, but it can also be caused by bacterial infections, toxic substances, or autoimmune disorders . Myocarditis is more common in younger patients, although it affects patients of all ages. Fulminant myocarditis, although rare, can result in life-threatening cardiogenic shock . Diagnosis of myocarditis is made using CMRI characterized by the presence of diffuse myocardial edema on T2 and with myocardial biopsy . In a meta-analysis of five observational studies with available CMRI data, one-third of MINOCA patients had myocarditis. It was more common in younger patients and those with high C-reactive protein .

ELIGIBILITY:
Inclusion Criteria:

* All patients; diagnosed with myocardial infarction with nonobstructive coronary arteries (MINOCA)
* clinical symptoms
* ECG : ischemic changes with or without ST segment elevation
* Echocardiograpy : segmental wall motion abnormalities (SWMA)
* positive cardiac enzymes
* Coronary angiography: insignificant lesions ,the absence of culprit obstructive coronary artery disease (epicardial coronary artery stenosis ≥50%)

Exclusion Criteria:

* Significant coronary artery disease (>50% stenosis) on angiography.
* Prior history of myocarditis or cardiomyopathy.
* Contraindications to CMR (e.g., pacemakers, severe renal dysfunction).

Ages: 17 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study Population Description Myocardial infarction patients who were underwent PPCI and the coronary angiography showing insignificant lesions (stenosis less than 50% )
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of myocarditis in patients presenting with MINOCA, as diagnosed by CMR. | 1 years
  Studying The incidence of myocarditis in MINOCA patients

CONTACTS AND LOCATIONS:
Overall Officials: Ayman khairy Mohamed Hassan, Principal Investigator — Cardiology department; Khaled Mohamed Abdullah Mohamed, Principal Investigator — Cardiology department

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC9132767/